CLINICAL TRIAL: NCT06241495
Title: The Effect of Aromatherapy on Anxiety, Difficulty in Providing a Semen Sample and Semen Parameters
Brief Title: Aromatherapy in Providing a Semen Sample
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Menekşe Nazlı AKER (Other)
Responsible Party: Sponsor-Investigator, Menekşe Nazlı AKER, Assist. Prof., Ankara University
Organization: Ankara University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: İ04-205-23
Record Dates: First submitted 2024-01-18; First posted 2024-02-05 (Actual); Last update posted 2025-02-12 (Actual); Status verified 2024-01

CONDITIONS: Infertility, Male
MeSH Terms: conditions — Infertility, Male | interventions — Aromatherapy

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Aromatherapy (Experimental)
  Interventions: Other: Aromatherapy
- Control Group (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Placebo — Placebo oil will be applied to the individuals included in the study. During the semen sample giving process, coconut oil (placebo) will be applied with a diffuser.
  Arms: Control Group
Other: Aromatherapy — Aromatherapy will be applied to the individuals included in the study. During the semen sample giving process, lavender oil will be applied with a diffuser.
  Arms: Aromatherapy

SUMMARY:
The aim of this study is to evaluate the effect of aromatherapy on the anxiety and difficulty of providing a semen sample and on semen volume, sperm concentration and motility percentage.

The study will be carried out in two different groups. After the men are evaluated in terms of eligibility criteria for the research, the men who are eligible will be informed about the research and written informed consent will be obtained from the men who accept. The random distribution of men to the study groups will be carried out random. The following applications will be made to the groups. Aromatherapy/placebo will be applied to the individuals included in the study. During the semen sample giving process, lavender oil/coconut oil (placebo) will be applied with a diffuser.

ELIGIBILITY:
Inclusion Criteria:

* Having applied to the center where the research will be conducted with a complaint of infertility
* Being 18 years or older

Exclusion Criteria:

* Individuals giving up on participating in the study
* Participant not being able to provide a semen sample
* Being diagnosed with azoospermia-oligozoospermia

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 102 (Actual)
Dates: Start 2024-01-29 (Actual); Primary Completion 2024-08-28 (Actual); Study Completion 2024-08-30 (Actual)

PRIMARY OUTCOMES:
Change in anxiety | before providing a semen sample, immediately after providing a semen sample
  The State-Trait Anxiety Inventory-S consist of 20 items with four points likert scales, each (not at all, somewhat, moderately so, very much so). Scores thus range between 20, indicating a low level of anxiety and 80, indicating a high level.
Anxiety about providing a semen sample | immediately after providing a semen sample
  VAS is a 10-cm-long measurement tool. The left end of the scale reads "no anxiety " and the right end reads "very anxious". A high score on the scale indicated a high level of anxiety and a score of 0 pointed to no anxiety.
Difficulty providing a semen sample | immediately after providing a semen sample
  VAS is a 10-cm-long measurement tool. The left end of the scale reads "not difficult" and the right end reads "very difficult ". A high score on the scale indicated a high level of difficulty and a score of 0 pointed to no difficulty.

SECONDARY OUTCOMES:
Semen volume | immediately after providing a semen sample
  Volume of semen sample
sperm concentration | immediately after providing a semen sample
  sperm concentration of semen sample
sperm motility percentage | immediately after providing a semen sample
  sperm motility percentage of semen sample
Total sperm count | immediately after providing a semen sample
  Total sperm count of semen sample
Satisfaction with the oil used | immediately after providing a semen sample
  VAS is a 10-cm-long measurement tool. The left end of the scale reads "I am not satisfied at all" and the right end reads "very satisfied". A high score on the scale indicated a high level of satisfied and a score of 0 pointed to no satisfied.

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara University Fertility Diagnosis, Treatment, Research and Application Center, Ankara, Turkey (Türkiye)